CLINICAL TRIAL: NCT06954389
Title: Hyperbaric Oxygen Therapy as a Neuroprotective Modality in Pediatric Acquired Brain Injury With Motor Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Eman Mohammed Abdel Hamid Gaml, Assistant Lecturer of Pediatrics, Faculty of Medicine, Kafr Elsheikh University, Kafr Elsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-137
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hyperbaric Oxygen Therapy; Neuroprotective; Pediatric; Acquired Brain Injury; Motor Disability
MeSH Terms: conditions — Brain Injuries | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric oxygen therapy group (Experimental): Patients received hyperbaric oxygen therapy using a monochamber hyperbaric chamber in addition to conventional rehabilitation.
  Interventions: Other: Hyperbaric oxygen therapy
- Control group (Active Comparator): Patients received conventional rehabilitation alone.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Hyperbaric oxygen therapy — Patients received hyperbaric oxygen therapy using a monochamber hyperbaric chamber in addition to conventional rehabilitation.
  Arms: Hyperbaric oxygen therapy group
Other: Conventional rehabilitation — Patients received conventional rehabilitation alone.
  Arms: Control group

SUMMARY:
This study aimed to assess the efficacy of hyperbaric oxygen therapy as a neuroprotective intervention in children with acquired brain injury.

DETAILED DESCRIPTION:
Pediatric acquired brain injury (ABI) represents a significant challenge in modern medicine, necessitating innovative therapeutic approaches to enhance recovery and minimize long-term neurological deficits.

Hyperbaric oxygen therapy (HBOT), which delivers oxygen at pressures exceeding atmospheric levels, has emerged as a promising neuroprotective intervention for various forms of pediatric brain injury, including traumatic brain injury (TBI), anoxic-ischaemic encephalopathy (AIE), and stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-12 years.
* Diagnosed with pediatric acquired brain injury confirmed by neurological examination and magnetic resonance imaging.
* Presence of neurological sequelae (e.g., cardiac arrest, intracranial hemorrhage, central nervous system infection, stroke, tumor, hypoxia).

Exclusion Criteria:

* Positive family history of degenerative brain insults.
* Behavioral problems.
* Contraindications to hyperbaric oxygen therapy :

  * Active epilepsy.
  * Respiratory insufficiency.
  * Uncontrolled heart failure.
  * Eustachian tube dysfunction.
  * Tympanic membrane rupture.
  * Mechanical ventilation dependency.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Spasticity assessment | Eight months post-intervention
  Spasticity assessment was conducted utilizing the Modified Ashworth Scale (MAS), which quantified resistance during passive soft tissue stretching.
  * Grade 0: No increase in muscle tone.
  * Grade 1: Slight increase in tone, minimal resistance.
  * Grade 2: More marked increase, resistance through most ROM.
  * Grade 3: Considerable increase, passive movement difficult.
  * Grade 4: Rigidity in flexion/extension.
  * Grade 5: Rigidity preventing passive movement.

SECONDARY OUTCOMES:
Evaluate changes in gross motor function temporally | Eight months post-intervention
  The Gross Motor Function Measure (GMFM) was utilized to evaluate changes in gross motor function temporally. This standardized assessment specifically quantified task completion capability rather than qualitative performance metrics.
  * Level I: Independent ambulation without limitations.
  * Level II: Walks without assistance but with limitations (e.g., uses handrails).
  * Level III: Walks with assistive devices (e.g., walker).
  * Level IV: Non-ambulatory but can move independently on hands and knees.
  * Level V: Complete dependence on a manual wheelchair for mobility.
Upper limb function assessment | Eight months post-intervention
  Upper limb function assessment (ULFA) was evaluated utilizing the Gordon and Duff Scale, which employed a six-point classification system (Types 0-5).
  * Type 0: No active upper extremity function.
  * Type 1: Minimal active movement, no functional use.
  * Type 2: Partial grasp and release, limited thumb opposition.
  * Type 3: Functional grasp but impaired precision tasks.
  * Type 4: Normal function with slight limitations (e.g., reduced speed).
  * Type 5: Normal or near-normal function with entire thumb opposition.
Assessment the fine motor function progression | Eight months post-intervention
  The Manual Ability Classification System (MACS) was implemented to assess fine motor function progression.
  * Level I: Handles objects easily and successfully.
  * Level II: Handles most objects with minor adaptations.
  * Level III: Handles objects with difficulty and requires assistance.
  * Level IV: Handles very few objects, highly dependent.
  * Level V: Does not handle objects and requires full support.
Evaluate feeding capabilities | Eight months post-intervention
  The Eating and Drinking Ability Classification System (EDACS) was employed to evaluate feeding capabilities.
  * Level I: Safe and efficient oral intake without assistance.
  * Level II: Minor dietary restrictions or compensatory strategies.
  * Level III: Moderate dietary restrictions and assistance.
  * Level IV: Requires alternative feeding methods (e.g., gastrostomy).
  * Level V: Complete dependence on non-oral feeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.